CLINICAL TRIAL: NCT05014971
Title: Multi-Stakeholder Engagement for Interdisciplinary Telehealth in Lewy Body Dementia
Brief Title: Telehealth in Lewy Body Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202001625; K23AG073575 (NIH); PRO00033145 (Other: UF UFIRST)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Lewy Body Dementia With Behavioral Disturbance; Lewy Body Parkinson Disease; Lewy Body Disease
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease

STUDY DESIGN:
Intervention Model Description: tele-neurohub model of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-neurohub (Experimental): This group will receive the tele-neurohub intervention which includes telemedicine appointments with the neurologist, speech therapist, social worker, and nutritionist at baseline, 3 months and 6 months, and PT and OT every 2 weeks for maintenance neuro-rehabilitation.
  Interventions: Behavioral: Tele-neurohub
- Usual care group (Active Comparator): Receive usual care but will have study visit assessments at baseline and 6 months.
  Interventions: Behavioral: Tele-neurohub

INTERVENTIONS:
Behavioral: Tele-neurohub — Interdisciplinary care delivered using telemedicine (zoom) technology which includes neurologist, physical, occupational and speech therapy, social worker and dietician.

SUMMARY:
Lewy body dementia (LBD) is the 2nd most common neurodegenerative dementia in the US. Optimal care requires an interdisciplinary approach, however often faced barriers include rural residence, limited access to specialists, travel distance, limited awareness of resources, and physical, cognitive, and behavioral impairments making travel to appointments challenging. Delivering interdisciplinary care remotely using video technology has the potential to improve access to care for patients with LBD.

DETAILED DESCRIPTION:
The purpose of this study is to convert an in-person patient-centric interdisciplinary care model to a virtual platform using stakeholder engagement from individuals with LBD, their caregivers and healthcare providers. Subsequently researchers will conduct a prospective, randomized, controlled pilot study implementing the virtual stakeholder developed interdisciplinary care model (tele-neurohub) for 6 month and assess the implementation outcomes of feasibility, acceptability, and appropriateness of the tele-neurohub model. The research goal is to establish and iteratively improve a virtual interdisciplinary model of care allowing patients with LBD and their caregivers to access sub-specialty care from their home.

ELIGIBILITY:
Participant with Lewy Body Dementia (LBD) Inclusion Criteria:

* LBD diagnosis by a dementia or movement disorders specialist
* Clinician-determined mild-moderate dementia severity
* Internet access with a Zoom-compatible device
* Caregiver who resides in the patient's home and is willing to participate
* Fluency in English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of completed tele-health visits | 6 months
  Feasibility will be determined by completion of at least 75% telehealth visits by the intervention cohort

SECONDARY OUTCOMES:
Satisfaction assessed by Patient Assessment of Communication of Telehealth questionnaire. | 6 months
  Acceptability will be determined by at least 80% of dyads reporting being "satisfied" or "highly satisfied" on the Patient Assessment of Communication of Telehealth questionnaire.
Appropriateness assessed by Intervention Appropriateness Measure | 6 months
  Appropriateness will be determined by the Intervention Appropriateness Measure, higher scores indicate greater appropriateness

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Patel, DO, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No